CLINICAL TRIAL: NCT00940238
Title: A Randomized, Single Dose, Open Label, Bioequivalence Study Comparing Citalopram Hydrobromide Tablets 40 mg (Torrent Pharmaceuticals Ltd) and RLD Tablets 40 mg (Manufactured By Forest Pharmaceuticals Inc, Missouri) in 24+2 Normal Healthy Male Subjects Under Fasting Condition
Brief Title: Study Comparing Citalopram Hydrobromide Tablets 40 mg (Torrent Pharmaceuticals Ltd) and RLD Tablets 40 mg (Manufactured By Forest Pharmaceuticals Inc, Missouri) in 24+2 Normal Healthy Male Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Torrent Pharmaceuticals Limited (Industry)
Other Study IDs: US/05/001
Record Dates: First submitted 2009-07-13; First posted 2009-07-15 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — Citalopram

INTERVENTIONS:
Drug: Citalopram Hydrobromide

SUMMARY:
* Objective:

  * To compare the rate and extent of absorption of Citalopram Hydrobromide Tablets 40 mg: Test Product: Citalopram Hydrobromide Tablets 40 mg manufactured by Torrent Pharmaceuticals Limited, India Reference Product: CelexaTM Tablets 40 mg (Reference Listed Drug) manufactured by Forest Pharmaceuticals Inc., Missouri under fasting conditions in 36 healthy, adult, human subjects in a randomized crossover study.
* Study Design:

  * Open-label, randomized, two period crossover studies in 36(Fasting)healthy, normal subjects to compare the single dose bioavailability of Torrent's Citalopram Hydrobromide tablets 40 mg and Forest Pharmaceutical's Celexa 40mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects in the range of 18 - 45 years of age.
* Body weight within ± 15% of the weight range as related to height, as per the Life Insurance Corporation (LIC) Chart (Appendix A).
* No abnormal findings as determined by baseline history, physical examination, vital signs (blood pressure, pulse rate, respiration rate and body temperature) hematological tests, serum chemistry, urinalysis, ECG and Chest X-ray. Subjects having values above/below the reference range, (Appendix J) for hematological, serum chemistry and urinanalysis values, will be clinically correlated for signs and symptoms. These subjects will be included if found asymptomatic.
* Willingness to follow, the protocol requirements, as evidenced by written, informed consent.
* Agreeing to, not to use any medication (prescription and over the counter), including vitamins and minerals for 15 days prior to study & during the course of the study.
* No history or presence of significant alcoholism or drug abuse in the past one year.
* Subjects should preferably be non-smokers. If moderate smokers are included (less than 10 cigarette per day) as per guidelines will be identified as such and documented in the history taking form in CRF.

Exclusion Criteria:

* Requiring medication for any ailment.
* Any medical or surgical conditions, which might significantly interfere with the functioning of gastrointestinal tract, blood-forming organs etc.
* History of cardiovascular, renal, hepatic, ophthalmic, pulmonary, neurological, metabolic or psychiatric diseases.
* Participation in a clinical drug study or Bioequivalence study 90 days prior to present study.
* History of malignancy or other serious diseases.
* Refusal to abstain from food for ten (10) hours prior to study drug administration on first day of each study period and for four (4) additional hours each, post dose.
* Refusal to abstain from water for one (1) hour prior to study drug administration on first day of each study period and for one (1) additional hour, post dosing.
* Any contraindication to blood sampling.
* Smoking or consumption of tobacco products during the study.
* Use of xanthine-containing beverages or food for 48 hours prior to each drug dose.
* Blood donation 30 days prior to the commencement of the study.
* Subjects with positive HIV tests.
* Subjects with positive HbsAg or Hepatitis-C tests.
* Known history of hypersensitivity Citalopram or related drugs.
* Pregnant and lactating women. At the time of screening, prior to enrollment, presence of pregnancy will be confirmed by urine pregnancy test.Just prior to commencement of study (for both periods), presence of pregnancy will be confirmed by urine pregnancy test.
* Female subjects not confirm to using birth control measures, from the date of screening till the completion of the second period of the study. Abstinence, barrier methods (condom, diaphragm, etc.) are acceptable. Use of hormonal contraceptives either oral or implants will not be acceptable.
* Female subjects whose menstruation cycle coincides with the study periods.
* History of drug abuse in the past one year.

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Accutest Research Laboratories Pvt. Ltd., Mumbai, Maharashtra, India